CLINICAL TRIAL: NCT00781469
Title: A Study to Evaluate the RNA Signature of Rheumatoid Arthritis From Synovium and Whole Blood
Status: Terminated | Type: Observational
Why Stopped: struggled to recruit and the synovial tissue samples obtained were so poor that we had to end the study prematurely without data from the primary outcomes
Sponsor: Imperial College London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 112009
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; RNA; Synovium; Peripheral blood mononuclear cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and synovium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Naive patients: 12 treatment naive patients who fulfil the American College of Rheumatology (ACR) criteria for RA with active disease defined by a Disease Activity Score (DAS)28 score of more than 3.2.
- Patients in remission: 6 RA patients in remission on a stable dose of methotrexate with a DAS28 score lower than 2.6
- Patients still have active disease: 12 patients who fulfill the ACR criteria for RA and are being treated with methotrexate but still have active disease, defined as a DAS28 score of more than 3.2

SUMMARY:
Rheumatoid arthritis is a systemic disease, it is not clear whether the gene expression profile exhibited by circulated peripheral blood cells and that expressed by the inflamed synovium mirror one another. Understanding this relationship would be useful not only in potentially having a relatively non-invasive means to predict response to therapy but it might be useful in better understanding differences in RA expression amongst patients with this disease, thus perhaps assisting in target identification through a better understanding of disease processes.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease affecting approximately 1% of the adult population. The disease is characterised by inflammation of synovial tissue (ST) in multiple joints, which often leads to destruction of joint integrity, contributing to serious functional impairment and disability. The contributors to its pathology include joint inflammation, abnormal cellular and humoral responses, and synovial hyperplasia. Ultrasonography is a powerful, non-invasive, and feasible way to evaluate synovial hyperplasia and guide its collection by biopsy.

ELIGIBILITY:
Inclusion criteria

* Adult men and non-pregnant, non-lactating women between 18 and 75 years of age. Sexually active females must be of either non-childbearing potential or willing to comply with the contraceptive requirements
* Body weight greater >40 kg and <120 kg with a body mass index (BMI) between 19-31 kg/m2
* Clinical history of rheumatoid arthritis as defined by ACR criteria
* Negative urine pregnancy test for women of child bearing age (except those with documented proof of hysterectomy or bilateral oophorectomy)

For populations B and C only

* Currently on a stable dosing regimen of methotrexate 7.5 to 25 mg once weekly, as their only DMARD (no changes in dosing regimen for 4 weeks prior to screening).

Exclusion criteria

* History of an acute illness within 2 weeks prior to the study
* History of drug abuse within 2 years
* Donation of blood in excess of 500 mL within 56 days prior to the first dose of study medication

For group A only

* Prior treatment with disease modifying anti-rheumatic agents or biologicals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and non-pregnant, non-lactating women between 18 and 75 years of age with a clinical history of rheumatoid arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Peripheral blood markers from patients with rheumatoid arthritis correlate to findings on ultrasound images and synovium (joint lining). | Initial visit

SECONDARY OUTCOMES:
Gene expression pattern of synovium in treatment naive rheumatoid arthritis patients correlates to that found in their circulating blood cells and if these are affected (or not)by disease modifying therapy (DMARD). | Visits 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Taylor, PhD, Principal Investigator — Imperial College London
Locations (1):
- Kennedy Institute Clinical Trials Unit, 4 West, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No